CLINICAL TRIAL: NCT03107546
Title: Comparison of Scar Formation in Syndactyly Release Surgery With Full Thickness Skin Graft Versus Skin Graft Substitute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gillette Children's Specialty Healthcare (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1703M09201
Record Dates: First submitted 2017-03-24; First posted 2017-04-11 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Syndactyly
Keywords: Syndactyly; Syndactyly release surgery; Full thickness skin graft; Hyalomatrix; Scar formation
MeSH Terms: conditions — Syndactyly | interventions — Skin Transplantation

STUDY DESIGN:
Intervention Model Description: Sample:
  The overall recruitment goal for the study is 40 participants within the first 5 years of the study.
  For phase one, a sample size of 10 participants is the goal, and the investigators anticipate that this will take at most 18 months to attain based on their historical data.
  For phase two, the investigators anticipate 30 months will be required to accumulate a sample size of 30 additional participants. Recruitment for phase two is expected to begin in year 2. Issues identified in the feasibility phase will be addressed as needed and the protocol amended.
Who Masked: Participant, Outcomes Assessor
Masking Description: The location of each (i.e., radial or ulnar side of the web) will be randomized and blinded. The participant and family will be blinded to which side of the web receives either the full-thickness graft or the skin substitute
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Skin graft (Other): full thickness skin graft
  Interventions: Other: Skin graft
- Hyalomatrix (Experimental): skin graft substitute
  Interventions: Device: Hyalomatrix

INTERVENTIONS:
Device: Hyalomatrix — We are comparing two techniques for covering the open area of the finger at the end of syndactyly release surgery. We would like to compare the current technique, a skin graft, with a new technique called Hyalomatrix.
  Arms: Hyalomatrix
Other: Skin graft — We are comparing two techniques for covering the open area of the finger at the end of syndactyly release surgery. We would like to compare the current technique, a skin graft, with a new technique called Hyalomatrix.
  Arms: Skin graft

SUMMARY:
Syndactyly is the most common hand abnormality in children. During development, two or more fingers do not separate in the usual way and remain connected by skin. Surgery is needed to separate the fingers. Usually, it is performed between 6 months and 3 years of age, depending on the severity of the syndactyly. During the surgery, the fingers are separated; however, there isn't enough skin to completely cover the fingers once they are separated. There are two areas on the fingers that need to be covered after separation, and there is a standard method, and now a new technique to cover these areas.

The standard current technique that surgeons use to cover the newly separated fingers is to apply a small section of the patient's own skin taken from a different area of their body (this is known as a skin graft).

A new technique called Hyaluronic acid matrix (Hyalomatrix®) is a U.S. Food and Drug Administration (FDA) approved, commercially available, skin graft substitute that is currently being used both in the US and in Europe. The Hyalomatrix (or skin graft substitute) is sutured into place using a stitch on each corner, over the areas left without skin covering during the surgery.

The purpose of this study is to compare effectiveness, wound healing, scar formation and potential associated complications of the current skin graft technique with the new technique called Hyalomatrix (or skin graft substitute) following surgery.

DETAILED DESCRIPTION:
Background/Significance:

Syndactyly is a congenital condition where children are born with webbing between their fingers. Syndactyly is the most common congenital hand condition in Caucasian children. Treatment for syndactyly is a syndactyly separation surgery, most commonly between 6 months and 3 years of age, depending on the severity of the syndactyly.

Syndactyly release surgery is typically performed by rearranging skin on the fingers and hand to cover the separated digits. However, there is seldom enough skin to cover all surfaces after separation of the digits and 2 similarly size defects are left, one at the base of each finger. The gold standard for covering these remaining defects has been full-thickness autograft skin. However, harvesting the graft, closing the defect at the harvest site and suturing the grafts into place requires considerable time (the investigators estimate a total of 60 minutes per web space). With recent concerns arising over prolonged anesthesia and brain development in young children, pediatric surgeons are searching for ways to limit anesthesia exposure. In addition to the prolonged anesthesia time for harvesting and suturing the autograft, the donor site is left with a scar that could be avoided if a skin graft substitute were available.

Hyaluronic acid matrix (Hyalomatrix®) is a FDA approved, commercially available, relatively inexpensive skin graft substitute. Each 1 inch by 1 inch sheet costs approximately $250.00 and could be used to cover both defects in most cases. It is sutured into place over a defect with a stitch on each corner. Although good results for use of HA matrix in syndactyly surgery have been reported in the European literature, no comparison has been made with the gold standard full thickness skin autograft.

Purpose:

The purpose of this study is to compare a Hyaluronic acid matrix skin graft substitute with full thickness autograft in the surgical treatment of syndactyly. While there are reports of successful use of this skin graft substitute for syndactyly surgery, it is important to compare any new treatment to the gold standard. The investigators wish to assess scar formation in syndactyly release surgery after use of a skin graft substitute (Hyalomatrix®) compared with the gold standard full-thickness skin graft. If the results with Hyalomatrix® are at least as good, or better, than full thickness skin graft, use of this skin graft substitute may significantly reduce surgical time, donor site morbidity, surgical suite expense, and anesthesia exposure to the developing brain.

Project Goals and Hypotheses:

The goal of this project is to compare the effectiveness of skin graft substitute (i.e., Hyalomatrix®) in syndactyly release surgery to the current gold standard full-thickness skin autograft. Utilization of a skin graft substitute following syndactyly surgery is presumed to be a safe and inexpensive method to promote wound healing, reduce scar formation, and consequently limit complications and scarring associated with skin autograft. Circumvention of the full-thickness skin graft not only decreases donor site morbidity, but is also expected to reduce the duration of surgery compared to using skin grafting alone, thus minimizing concerns associated with prolonged sedation in children. Currently, a single web syndactyly release takes approximately 2 hours, with approximately 1 hour of time for graft harvest and placement.

The investigators hypothesize that there is no significant difference in scaring; healing and scar formation between the FDA approved skin graft substitute, Hyalomatrix®, and the gold standard full-thickness skin graft when used during syndactyly release surgery. This will be measured by comparing scores (on the Patient/Parent and Observer Scar Assessment (POSAS), the modified Hamilton burn scar rating by photographic analysis and the Web Creep Assessment) of the sites with full-thickness skin graft versus sites with Hyalomatrix. These measurement tools assess the thickness, color (darkness), pliability, appearance, and vascularity (redness) of a scar compared to normal skin and includes assessments by both provider and participant (parent).

Study Design and Methodology:

A randomized, single-blinded, within-subject controlled study will be performed to compare the effectiveness of skin graft substitute to the gold standard full-thickness skin autografts for children requiring syndactyly release surgery. The study will have two phases. Phase one will serve as a feasibility study and will include n=10 children undergoing surgical intervention for one, or more, syndactylized webs on their hand(s). Phase one will serve as a feasibility study to conduct power analysis, potential adverse events and identify issues in the protocol. The investigators do not have any specific safety concerns, as Hyalomatrix is FDA approved for use in children. However, the investigators do not have personal experience in its use. Preliminary analyses will be done after initial inclusion of 10 webs, or approximately 5 children and again following the inclusion of all 10 children in phase one. Phase two will implement improvements identified in phase 1, and will include n=30 new participants.

In both phases, the participants and caregiver(s) will remain as blinded as possible to the specific location of the full-thickness skin graft and skin graft substitute (i.e., radial or ulnar side of the syndactyly-released web) until after the study has been completed. The provider removing the bandage will attempt to remove the silicone sheet from the Hyalomatrix site with the postop dressing. Thus each web will have an internal control, or gold-standard graft. This within-subject comparison is expected to minimize variability in intra- and inter-patient healing irregularities, as well as intra- and inter-surgeon performance and therefore provide a more valid comparison of the equivalency of the two techniques.

Participants will be followed clinically, per standard of care, with the exception of long-term follow up (i.e., 24 month post-surgery assessments), in which parents will be asked to answer a set of questions online via a secure data collection tool called REDCap. Informed consent will be obtained from parent(s) or legal guardian(s) for children under the age of 18 year old. Written assent will be obtained from study participants between the ages of 8 years old through 16 years old. For participants who are 8 and older and unable to sign the assent form, verbal consent will be documented on the assent form by the person leading the consent process.

Participants, caregivers and providers will regularly complete the outcome measures below, at the treating surgeons' post-surgical standard of care follow-up visit schedule. Standard of care visits typically occur 0-4 weeks, and approximately at 8 weeks, 6 months, 12 months and 24 months post-surgery. Scheduled completion of outcome measures is denoted below. Please note, the first post-operative visit is intended to remove the initial cast which may or may not require recasting. Due to variability in patient care, outcome measure for the study will not be collected beyond photographs and documenting any adverse events.

Interventions:

For consented and enrolled participants, each web that requires surgical-intervention will receive both a skin graft substitute (Hyalomatrix®) and a full-thickness skin autograft. The location of each (i.e., radial or ulnar side of the web) will be randomized and blinded. The participant and family will be blinded to which side of the web receives either the full-thickness graft or the skin substitute. The skin substitute will be sutured into place with standard absorbable sutures at the corners of the skin substitute. The skin substitute will overlap the edges of the normal skin by a few millimeters. At the three week visit, the Hand Service Nurse, surgeon, or trained staff will personally remove the cast of all participants enrolled in the study, along with the Hyalomatrix® backing (visible layer not present on the full-thickness graft, which may unblind the family), prior to the family seeing the wound. This precaution is intended to keep the family blinded to the specific location of the graft substitute.

Upon completion of the study at 24 months post-surgery, parents will first be asked to self-identify the location of the gold-standard vs the skin graft substitute for each web, and both the parents and observers will complete a satisfaction/preference questionnaire, followed by formal unbinding via a letter. For participants who prematurely discontinue their participation prior to the conclusion of the study, the same unblinding letter will be sent the home revealing the location of the skin graft substitute and traditional graft.

Surgery:

REDCap will be used for the randomization of each web requiring surgical release. Specifically, for each web undergoing surgery, REDCap will assign the specific location (i.e., radial and ulnar side of each of the surgically released web) that the skin substitute and full-thickness skin graft are to be placed for each of the webs. Consequently, one side of a single web will have the gold-standard full-thickness skin autograft (i.e., control side of the web), and the other side will have the skin substitute.

Secondary outcome measures:

Secondary outcome measures include, participants' demographics, clinic visit information including radiographs, and surgery related measures. A satisfaction questionnaire will also be given to participants/families and observers at the end of the study to assess preferred grafted side (Hyalomatrix® vs full-thickness graft), equivalency of the two graft sites and donor scar, and surgical technique (for the observer only). These outcomes will be used in sub analyses or co-variates for the primary outcome measures.

Data Analysis:

For statistical analyses, the sample size will utilize matched-pairs of surgically operated webs (i.e., full-thickness skin graft versus Hyalomatrix®), rather than participants. It is expected that the sample size of webs will exceed the number of participants enrolled in the study (i.e., n=40 participants may result in approximately 60 webs). Preliminary statistical analyses will be performed at the conclusion of phase one, and will determine whether the sample size of n=30 participants provides sufficient statistical power.

The effectiveness of skin graft substitute (i.e., Hyalomatrix®) in syndactyly release surgery compared to the current gold standard full-thickness skin autograft will be assessed by comparing the Patient Scar Assessment Scores, Observer Scar Assessment Scores, Hamilton scores and web creep for each web. The summated total scores of these tools will be compared using Wilcoxon Signed Rank tests with a matched pair (hyalomatrix vs full-thickness graft) design over time (8 weeks, 6 months, 12 months and 24 months post-surgery).

Descriptive statistics will be used to describe participant demographics, clinic visit information, adverse events, and satisfaction surveys at the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients under the age of 18 years who require syndactyly release surgery with skin grafting for one, or more, web spaces on their hand(s) will be eligible for this study
2. Those who have had a previous syndactyly release surgery on one or more webs will still be considered for inclusion if the current web requiring syndactyly surgery has not been previously operated on

Exclusion Criteria:

1. Previous surgery on the web that requires a subsequent syndactyly release
2. Diagnosis of macrodactyly
3. Those who otherwise do not meet the inclusion criteria

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in scar quality between Hyalomatrix® and full-thickness skin graft when used during syndactyly release surgery as assessed by the Patient/Parent and Observer Scar Assessment Scale (POSAS) and the Hamilton Photographic Scar Assessment Scale | 24 months
  The difference in scar quality between Hyalomatrix and full thickness skin graft will be assessed by the POSAS and the Hamilton Photographic Scar Assessment Scales at 8 weeks, 6 months, 12 months and 24 months after surgery. These scales assess the thickness, color (darkness), pliability, appearance, and vascularity (redness) of a scar compared to normal skin and includes assessments by both the investigators and participant/caregiver. Wilcoxon signed-rank tests will be utilized to compare total scores for the Hyalomatrix and the full-thickness skin graft as matched pairs over time.
Difference in web creeping between Hyalomatrix® and full-thickness skin graft when used during syndactyly release surgery as assessed by the Web Creep Assessment Scale. | 24 months
  The difference in web creeping between Hyalomatrix and full thickness skin graft will be assessed by the Web Creep Assessment Scale. This scale will be assessed by the investigators using photographs of the participant's hands. Photographs will be taken at immediately pre-surgery, immediate post-surgery, 8 weeks, 6 months, 12 months and 24 months. Wilcoxon signed-rank tests will be utilized to compare total scores for the Hyalomatrix and the full-thickness skin graft as matched pairs over time.

SECONDARY OUTCOMES:
Analysis of the participants' demographic, clinical and surgical data to see if there is any difference between the Hyalomatrix® and full-thickness skin graft groups. | 24 months
  Descriptive statistics will be used to analyze the participants' demographic, clinical and surgical data.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Van Heest, MD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States

REFERENCES:
- [Background] Dao KD, Wood VE, Billings A. Treatment of syndactyly. Tech Hand Up Extrem Surg. 1998 Sep;2(3):166-77. doi: 10.1097/00130911-199809000-00004. No abstract available. PMID 16801754
- [Background] Perna RB, Loughan AR, Le JA, Hertza J. Prenatal and perinatal anesthesia and the long-term cognitive sequelae: a review. Appl Neuropsychol Child. 2015;4(1):65-71. doi: 10.1080/21622965.2013.779275. Epub 2013 Oct 24. PMID 24156239
- [Background] Landi A, Garagnani L, Leti Acciaro A, Lando M, Ozben H, Gagliano MC. Hyaluronic acid scaffold for skin defects in congenital syndactyly release surgery: a novel technique based on the regenerative model. J Hand Surg Eur Vol. 2014 Nov;39(9):994-1000. doi: 10.1177/1753193414529046. Epub 2014 Mar 24. PMID 24664163
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Crowe JM, Simpson K, Johnson W, Allen J. Reliability of photographic analysis in determining change in scar appearance. J Burn Care Rehabil. 1998 Mar-Apr;19(2):183-6. doi: 10.1097/00004630-199803000-00019. PMID 9556325
- [Background] Withey SJ, Kangesu T, Carver N, Sommerlad BC. The open finger technique for the release of syndactyly. J Hand Surg Br. 2001 Feb;26(1):4-7. doi: 10.1054/jhsb.2000.0575. PMID 11162004

DOCUMENTS (1):
  • Informed Consent Form (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT03107546/ICF_000.pdf